CLINICAL TRIAL: NCT00029965
Title: Natural History of Glycosphingolipid Storage Disorders and Glycoprotein Disorders
Status: Recruiting | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020107; 02-HG-0107
Record Dates: First submitted 2002-01-27; First posted 2002-01-28 (Estimated); Last update posted 2026-01-15 (Actual); Status verified 2026-01-05

CONDITIONS: Neurological Regression; Myoclonus; Cherry Red Spot; Brain Atrophy
Keywords: Sialidosis; Lysosomal Storage; GM1 Gangliosidosis; GM2 Gangliosidosis; Natural History; Glycoprotein Disorders; Lysosomal Storage Disorder; Tay-Sachs; Sandhoff; Gaucher
MeSH Terms: conditions — Myoclonus; Mucolipidoses; Gangliosidosis, GM1; Gangliosidoses, GM2; Lysosomal Storage Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Glycoprotein Disorders: Glycoprotein Disorders
- Lysosomal Storage Diseases: Lysosomal Storage Diseases

SUMMARY:
Study description:

This is a natural history study that will evaluate any patient with enzyme or DNA confirmed GM1 or GM2 gangliosidosis, sialidosis or galactosialidosis. Patients may be evaluated every 6 months for infantile onset disease, yearly for juvenile onset and approximately every two years for adult-onset disease as long as they are clinically stable to travel. Data will be evaluated serially for each patient, and cross-sectionally for patients of similar ages and genotypes. Genotype-phenotype correlations will be made where possible although these are rare disorders and the majority of the patients are compound heterozygotes.

Objectives:

To study the natural history and progression of neurodegeneration in individuals with glycosphingolipid storage disorders (GSL), GM1 and GM2 gangliosidosis, and glycoprotein (GP) disorders including sialidosis and galactosialidosis using clinical evaluation of patients and patient/parent surveys.

To develop sensitive tools for monitoring disease progression.

To identify biological markers in blood, cerebrospinal fluid, and urine that correlate with disease severity and progression and can be used as outcome measures for future clinical trials.

To further understand and characterize the mechanisms of neurodegeneration in GSL and GP storage disorders across the spectrum of disease beginning with ganglioside storage in fetal life.

Endpoints:

Exploring the natural history of Lysosomal Storage Diseases and Glycoprotein Disorders

Study Population:

Patients with enzyme or DNA confirmed GM1 or GM2 gangliosidosis, sialidosis or galactosialidosis. Accrual ceiling is 200 participants. No exclusions based on age, gender, demographic group, or demographic location. Patients included in our study are those that are seen at the NIH Clinical Center, subjects that have only sent in blood samples, as well as those who complete the questionnaire or provided head circumference measures.

DETAILED DESCRIPTION:
The GM1 and GM2 gangliosidoses are rare lysosomal storage disorders that primarily affect the brain and are uniformly fatal. The glycoproteinoses sialidosis and galactosialidosis are ultra-rare disorders involving predominantly the skeletal and central nervous systems that are likewise fatal or severely debilitating. No effective therapy for patients with these diseases has yet been demonstrated. Historically, since these disorders are fatal very little natural history information or disease characterization using modern medical techniques has been collected. This information is vital to establish the pattern of disease progression and to identify clinical, biochemical and biophysical markers that can be used as endpoints in future therapeutic trials.

This protocol aims to study the natural history of the GM1 and GM2 gangliosidoses, sialidosis and galactosialidosis in affected individuals of all ages, races and genders using medical technologies including MRI/MRS, hearing evaluation and auditory evoked response testing, EEG, sleep study, EMG/NCV, echocardiogram and abdominal ultrasound as well as subspecialty evaluations in rehabilitative medicine (including gait analysis), ophthalmology, speech language pathology, neurology, and psychology. Biomarkers of disease progression may be explored in CSF, blood, and urine samples for correlation with disease staging. Fibroblast cultures will be established for testing potential therapeutic agents. Some fibroblast lines will be used to create induced pluripotent stem cells (iPSC) for differentiation into neural tissues, more relevant for the study of these disorders that primarily affect the central nervous system (CNS). We hypothesize that relevant biomarkers will correlate with disease progression and will shed light on the pathophysiology of disease progression in these devastating disorders.

As a means of acquiring additional information, subjects or their parents may also be asked to complete a questionnaire regarding their medical and developmental history, initial clinical presentation of the disease and steps toward diagnosis. At their request, the same questionnaire may be sent to families who do not wish to undergo clinical evaluation at the NIH, who are medically fragile and unable to travel, or whose affected member(s) are already deceased.

We know that children with infantile GM2 gangliosidosis develop increasing macrocephaly as part of their disease. No "normal" curves for head circumference vs. age currently exist for this disorder. In an attempt to provide such curves to the clinical community parents may also be asked to provide head circumference data on their children whether they are being seen at NIH or whether a clinical questionnaire is being completed for children too medically fragile to travel or already deceased.

We know that for infantile onset disease the storage of ganglioside in neurons begins during the second trimester of pregnancy. In rare situations where carrier couples learned from prenatal diagnosis that they were carrying a fetus with infantile disease and had decided to terminate the pregnancy, we accepted samples of fetal tissue prior to June 5, 2019, for analysis of biomarkers including gene expression analysis that may lend clues as to the underlying pathogenesis of disease. This may lead to increased understanding of the early events in disease pathogenesis and suggest possible therapies.

We anticipate that information obtained from the small population of patients with glycosphingolipid and glycoprotein disorders evaluated in this study will have a broader impact on patients with other neurodegenerative lysosomal storage disorders and perhaps more common disorders of neurodegeneration.

ELIGIBILITY:
* INCLUSION CRITERIA:

Any individual with GM1 or GM2 gangliosidosis, sialidosis or galactosialidosis documented by enzyme deficiency or mutation analysis in a CLIA-approved laboratory will be eligible for the study.

EXCLUSION CRITERIA:

There will be no exclusion based on race, gender, or ethnicity; however particular ethnic groups may be overrepresented due to the frequency of the diseases in a specific population (e.g., Ashkenazi Jews in infantile and adult GM2 and Roma "travelers" in juvenile GM1). The majority of juvenile subjects will have severely impaired decision-making and even informed assent in older children may not be possible. Children with Morquio B disease are not expected to be cognitively impaired. The children with Morquio B ages 7-11 years will be asked to give verbal assent and ages 12-17 years will be asked to give written assent to the protocol. Some subjects who have reached the age of 18 may need to have legally authorized representative (usually their parents) sign consent on their behalf.

Ages: 1 Day to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Lysosomal Storage Diseases and Glycoprotein Disorders.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2002-02-06 (Actual)

PRIMARY OUTCOMES:
Exploring the natural history of Glycoprotein Disorders | Assessed one to every two years
  Exploring the natural history of Glycoprotein Disorders
Natural history of Lysosomal Storage Diseases | Assessed one to every two years
  Exploring the natural history of Lysosomal Storage Diseases

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia J Tifft, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
There is not currently a plan to make IPD available, however, after publishing trial data, a plan to share IPD may be made.

REFERENCES:
- [Background] Wada R, Tifft CJ, Proia RL. Microglial activation precedes acute neurodegeneration in Sandhoff disease and is suppressed by bone marrow transplantation. Proc Natl Acad Sci U S A. 2000 Sep 26;97(20):10954-9. doi: 10.1073/pnas.97.20.10954. PMID 11005868
- [Background] Cantor RM, Roy C, Lim JS, Kaback MM. Sandhoff disease heterozygote detection: a component of population screening for Tay-Sachs disease carriers. II. Sandhoff disease gene frequencies in American Jewish and non-Jewish populations. Am J Hum Genet. 1987 Jul;41(1):16-26. PMID 2955697
- [Background] Myerowitz R, Hogikyan ND. Different mutations in Ashkenazi Jewish and non-Jewish French Canadians with Tay-Sachs disease. Science. 1986 Jun 27;232(4758):1646-8. doi: 10.1126/science.3754980.
- [Derived] Han ST, Hirt A, Nicoli ER, Kono M, Toro C, Proia RL, Tifft CJ. Gene expression changes in Tay-Sachs disease begin early in fetal brain development. J Inherit Metab Dis. 2023 Jul;46(4):687-694. doi: 10.1002/jimd.12596. Epub 2023 Feb 5. PMID 36700853
- [Derived] Luckett A, Yousef M, Tifft C, Jenkins K, Smith A, Munoz A, Quimby R, Porter FD, Dang Do AN. Anesthesia outcomes in lysosomal disorders: CLN3 and GM1 gangliosidosis. Am J Med Genet A. 2023 Mar;191(3):711-717. doi: 10.1002/ajmg.a.63064. Epub 2022 Dec 2. PMID 36461157
- [Derived] Daich Varela M, Zein WM, Toro C, Groden C, Johnston J, Huryn LA, d'Azzo A, Tifft CJ, FitzGibbon EJ. A sialidosis type I cohort and a quantitative approach to multimodal ophthalmic imaging of the macular cherry-red spot. Br J Ophthalmol. 2021 Jun;105(6):838-843. doi: 10.1136/bjophthalmol-2020-316826. Epub 2020 Aug 4. PMID 32753397
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2002-HG-0107.html